CLINICAL TRIAL: NCT01070446
Title: Choline Nutrition in Children With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Dr. Sheila M. Innis, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H06-7044
Record Dates: First submitted 2010-02-10; First posted 2010-02-18 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Cystic Fibrosis
Keywords: choline; cystic fibrosis; methyl metabolism; fatty acids; oxidative stress; pulmonary function
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): This study involves children with CF who will take a water soluble vitamin supplement of choline bitartrate, 2 gm per day with meals.
  Interventions: Dietary Supplement: Vitamin: Choline Bitartrate (2-hydroxyethyl) trimethylammonium salt 1:1

INTERVENTIONS:
Dietary Supplement: Vitamin: Choline Bitartrate (2-hydroxyethyl) trimethylammonium salt 1:1 — This is a prospective, repeated measures study involving children with Cystic Fibrosis. Children will be assessed (1) before starting the choline supplement, (2) after taking the supplement for 6 months and after the supplement has been discontinued for 3 months.

SUMMARY:
Cystic fibrosis (CF) is the most common lethal, inherited disorder among Caucasians. Choline is an essential vitamin and as a methyl donor is critically needed to support the normal metabolism. Our previous studies have demonstrated that children with CF have depleted levels of choline. The purpose of this study is to supply a choline supplement to children with CF to see if their nutrition and methyl status can be improved.

DETAILED DESCRIPTION:
This will be a prospective, repeated measures study involving 34 children with CF who will take a supplement of water soluble choline bitartrate, 2 gm/day with meals for 6 months. The baseline (day 0) results for each child will serve as his/her own control, and assessments will be made at 3 months and 6 months choline supplementation and again 3 months after stopping choline.

The supplement will be provided as capsules containing 250 mg choline bitartrate. 4 capsules will be taken with or immediately before each of two meals per day: breakfast and dinnertime meals, providing 1 gm of supplemental choline each day.

The children will be enrolled by description of the project to the child and their parent(s) at a CF clinic appointment. Body weight, height and blood pressure will be measured and routine blood work including liver enzymes, hematology, serum zinc, selenium and vitamins A and E will be completed as part of the clinic appointment. The hematology and clinical chemistry will be done by the Hematopathology and Clinical Chemistry labs at the B.C.'s Children's Hospital. CF genotype, gender, birth date, hematology, clinical chemistry, anthropometry, nutritional measures, pulmonary function test results, chest X-Ray and/or CT scans, pancreatic function test results (fecal elastase, chymotrypsin or secretin-CCK), medications and supplements (including enzymes, vitamins, minerals, nutrition supplements & Natural Health Products) and where available, liver ultrasound and biopsy reports will be collected from chart data. Information in the subject's medical charts relating to antibiotic therapy, duration of illnesses, hospitalization and diagnosis will be reviewed to ensure the inclusion/exclusion criteria are met.

Assessment of pulmonary function by computer assisted spirometry which includes the measures of forced vital capacity (FVC), forced expiratory volume in one second (FEV1) and forced mid-expiratory flow (FEF 25-75) is completed for all children as part of each regularly scheduled clinic visit and the results collected for this study.

ELIGIBILITY:
Inclusion Criteria:

* children aged 5-17 yr with proven CF and known genotype
* with stable pulmonary disease, are outpatients with no hospitalizations or changes to antibiotic regiment during the previous 1 month and not receiving any parenteral nutrition
* are non-smokers without asthma, may be taking routine fat soluble vitamins but must not be taking any supplemental fish oil, docosahexanoic acid (DHA) or choline containing compounds, experimental drugs or any aerosol or oral interventions designed to deliver or increase glutathione or receiving oral or parenteral corticosteroidal medications. E.g prednisone.

Exclusion Criteria:

* are not 5-17 years of age, do not have CF or have the medical condition trimethylaminuria.
* have CF, but have allergies to any of the ingredients in the choline supplements; are hospitalized; have asthma or are smokers; are taking oral or parenteral corticosteroidal medications or any intravenous nutritional support; have kidney or liver disease; or have a baseline FEV 1 of less than 50% predicted value (which at our clinic means they are likely hospitalized or about to be admitted to hospital).

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
plasma choline, SAM, SAM/SAH ratio, homocysteine, GSH and the GSH/GSSG | 9 months

SECONDARY OUTCOMES:
(2-hydroxyethyl) trimethylammonium salt (1:1) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M. Innis, Dr., Principal Investigator — University of British Columbia
Locations (1):
- Child & Family Research Institute, CF Clinic, Vancouver, British Columbia, Canada